CLINICAL TRIAL: NCT02569957
Title: Evaluation of the Addition of N-Acetylcysteine to Topotecan in the Tumor Microenvironment of Persistent or Recurrent High Grade Endometrioid or Serous Ovarian Carcinoma
Brief Title: Effect of Acetylcysteine With Topotecan Hydrochloride on the Tumor Microenvironment in Patients With Persistent or Recurrent High Grade Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was halted prematurely due to slow accrual.
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15P.404; JT 7408 (Other: JeffTrial Number)
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Malignant Ovarian Endometrioid Tumor; Malignant Ovarian Serous Tumor; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Topotecan; Acetylcysteine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (topotecan hydrochloride) (Active Comparator): Patients receive topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15 (+/- 1 day window for each treatment day). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Topotecan Hydrochloride
- Arm II (topotecan hydrochloride, acetylcysteine) (Experimental): Patients receive topotecan hydrochloride as in Arm I. Patients also receive acetylcysteine IV over 60 minutes on days 1, 8, 15, and 22 (+/- 1 day window for each treatment day) and acetylcysteine PO BID on days 2-7, 9-14, 16-21, and 23-28, unless administration window was utilized. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Topotecan Hydrochloride; Drug: Acetylcysteine

INTERVENTIONS:
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamtin
  Arms: Arm I (topotecan hydrochloride)
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamtin
  Arms: Arm II (topotecan hydrochloride, acetylcysteine)
Drug: Acetylcysteine — Given IV and PO
  Other Names: N-acetylcysteine; N-acetyl-L-cysteine (NAC)
  Arms: Arm II (topotecan hydrochloride, acetylcysteine)

SUMMARY:
This randomized phase II trial studies the effects of acetylcysteine and topotecan hydrochloride on the tumor microenvironment, or cells that make up a tumor, compared to topotecan hydrochloride alone in patients with ovarian, fallopian tube, or primary peritoneal cancer that has not responded to treatment (persistent) or has returned after a period of improvement (recurrent) and is high grade (likely to grow and spread quickly). Research has shown that cancer cells may be able to convert nearby normal cells into cancer cells. Acetylcysteine may stop this from happening. Topotecan hydrochloride is a chemotherapy drug used to treat ovarian cancer, and may help acetylcysteine work better. This trial studies the effect of acetylcysteine and topotecan hydrochloride on the tumor microenvironment to see if they can help make it more difficult for tumor cells to grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of subjects with persistent or recurrent high grade endometrioid or serous ovarian carcinoma who demonstrate a downregulation of monocarboxylate transporter 4 (MCT4) in the ovarian stroma in response to exposure to topotecan (topotecan hydrochloride) and N-acetylcysteine (NAC) (acetylcysteine) as compared to topotecan alone.

SECONDARY OBJECTIVES:

I. To determine the expression levels of caveolin 1 (Cav-1), solute carrier family 16 (monocarboxylate transporter), member 1 (MCT1), translocase of outer mitochondrial membrane 20 homolog (yeast) (TOMM20), fatty acid binding protein 4, adipocyte (FABP4), hypoxia inducible factor 1, alpha subunit (HIF-1 alpha) and NF kappaB activating protein (NFκB) in pathological samples of tumors after therapy with NAC relative to samples taken at time of initial diagnosis.

II. To assess the potential impact of NAC on progression free survival, overall survival, objective tumor response- complete or partial, and duration of response.

III. To estimate the proportion of subjects who survive progression free for at least 6 months and the proportion of patients who have objective tumor response, complete or partial in response to therapy IV. To assess safety and tolerability of NAC plus topotecan treatment in subjects with endometrioid or serous ovarian carcinoma by Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0 criteria.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive topotecan hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15 (+/- 1 day window for each treatment day). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive topotecan hydrochloride as in Arm I. Patients also receive acetylcysteine IV over 60 minutes on days 1, 8, 15, and 22 (+/- 1 day window for each treatment day) and acetylcysteine orally (PO) twice daily (BID) on days 2-7, 9-14, 16-21, and 23-28, unless administration window was utilized. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have persistent or recurrent high grade endometrioid or serous ovarian, primary peritoneal or fallopian tube carcinoma. Histologic documentation of the original primary tumor is required via the pathology report.
2. All patients must have measurable disease that is amenable to biopsy. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥20 mm when measured by conventional techniques including palpation, plain film x-ray, CT, and MRI, or ≥ 10 mm when measured by high resolution CT.
3. Patient must have at least one target lesion to be used to assess response on this protocol as defined by RECIST 1.1. Tumors within a previously irradiated field will be designated as non-target lesions unless progression is documented or a biopsy is obtained to confirm persistent disease at least 90 days following completion of radiation therapy.
4. Patients must have a GOG performance status of 0, 1, or 2.
5. Patients must be free of active infections requiring antibiotics, with the exception of uncomplicated urinary tract infections (UTIs).
6. Any hormonal therapy directed at the tumor must be discontinued at least one week prior to initiation of therapy. Continuation of hormone replacement therapies is permitted.
7. Any other prior therapy directed at the tumor, including immunologic agents, must be discontinued at least 3 weeks prior to initiation of therapy.
8. Patients must have had at least one prior platinum/taxane combination chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatin compound. This initial treatment may include intraperitoneal therapy, high dose therapy, consolidation, noncytotoxic agents, or extended therapy.
9. Patients must be platinum resistant- defined as progressive disease while receiving platinum therapy or within 6 months of completing first line platinum therapy or patients who have progressive disease after two lines of platinum based treatment.

   1. Cytotoxic regimens are any that include agents that target the genetic and/or mitotic apparatus of the dividing cells, resulting in dose limiting toxicity to the bone marrow or gastrointestinal mucosa
   2. Patients are allowed to receive, but not required to receive biologic (noncytotoxic) therapy as part of their treatment regimen, e.g. bevacizumab.
10. Patients Must Have Adequate:

    1. Bone Marrow Function: Absolute Neutrophil Count greater than or equal to 1000/mcl. Platelets greater than or equal to 100,000/mcl. Hemoglobin greater than 10 g/dl. (Patients may be transfused to achieve this hemoglobin.)
    2. Renal Function: creatinine less than or equal to 1.5 x upper limit of normal, CTCAE v 4.0 grade 1.
    3. Hepatic Function: bilirubin less than or equal to 1.5 x upper limit of normal, CTCAE v 4.0 grade 1. Asparate transaminase (AST) and alkaline phosphatase less than or equal to 2.5 x upper limit of normal, CTCAE v 4.0 grade 1.
    4. Coagulation: PT, PTT less than or equal to 1 to 1.5 x upper limit of normal CTCAE v 4.0 grade 1 except for patients on therapeutic anticoagulation.
    5. Neurologic Function: neuropathy (sensory and motor) less than or equal to CTCAE v 4.0 grade 1.
11. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
12. Patients must meet pre-entry requirements as specified.
13. In the unlikely event that patients are still of childbearing potential, these patients must have a negative serum pregnancy test within 72 hours prior to initiating protocol therapy and be practicing an effective form of contraception during protocol therapy and for at least 4 weeks following completion of protocol therapy.
14. Patients must be 18 years of age or older.
15. Patients must not be receiving any other investigational agent.
16. Patients must be able to swallow whole pills. -

Exclusion Criteria:

1. Patients who have had previous treatment with topotecan.
2. Patients who have had more than 4 prior chemotherapy regimens.
3. Patients who have received radiation to more than 25% of marrow-bearing areas.
4. Patients with a history of other invasive malignancies are excluded if there is any evidence of other malignancy being present within the last 3 years.
5. Patients who have received prior chemotherapy for any abdominal or pelvic tumor other than for treatment of ovarian carcinoma within the last 3 years are excluded. Patients may have received prior chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration and the patient remains free of recurrent of metastatic disease.
6. Pregnant or nursing women or women of childbearing potential unless using effective contraception as determined by the investigator. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2017-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schilder, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Demonstrate a Downregulation of MCT4
Description: The two-sided Fisher's exact test with alpha 0.05 will be used to compare the proportions of subjects who demonstrate a downregulation of MCT4 between subjects treated with topotecan hydrochloride and NAC and topotecan hydrochloride alone.
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Expression Levels of Cav-1 in Tissue Samples
Description: Evaluated in a generalized linear mixed effects model adjusting for the random subject effects. The expression levels will be log or otherwise transformed, if necessary, to satisfy the normal distribution assumption of the model. The fitted model will be used to evaluate the post-treatment change in the expression levels.
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Expression Levels of MCT1 in Tissue Samples
Description: as for outcome 2
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Expression Levels of TOMM20 in Tissue Samples
Description: as for outcome 2
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Expression Levels of FABP4 in Tissue Samples
Description: as for outcome 2
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Expression Levels of HIF-1 Alpha in Tissue Samples
Description: as for outcome 2
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Expression Levels of NFκB in Tissue Samples
Description: as for outcome 2
Time Frame: Baseline to up to day 20 after first course of topotecan hydrochloride
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Number of Circulating Tumor Cells
Description: Compared pre-therapy and post- 1 cycle of therapy with a Fisher's exact test.
Time Frame: Baseline to day 29
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Progression-free Survival
Description: Compared between the two arms using the log-rank test.
Time Frame: Up to 24 months
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Overall Survival
Description: Compared between the two arms using the log-rank test.
Time Frame: Up to 24 months
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Objective Tumor Response Rates
Description: Evaluated using the exact binomial confidence intervals and compared between the two arms using the Fisher's exact test.
Time Frame: Up to 24 months
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Duration of Response
Description: Compared between the two arms using the two-sample Wilcoxon test.
Time Frame: Up to 24 months
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Proportion of Patients Experiencing Adverse Events, Evaluated Using the National Cancer Institute CTCAE Version 4.0
Description: Tabulated and reported with the corresponding exact binomial confidence intervals.
Time Frame: Up to 24 months
Population: The trial was halted prematurely due to slow accrual. Data were not collected and the Outcome will never be analyzed.
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Arm I (Topotecan Hydrochloride) | Arm II (Topotecan Hydrochloride, Acetylcysteine)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Topotecan Hydrochloride) (N=0) | Arm II (Topotecan Hydrochloride, Acetylcysteine) (N=1)
Activated Partial Thromboplastin Time prolonged (Blood and lymphatic system disorders) | 0 (0) | 1 (9)
ANC decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatine Increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (8)
Dizziness (General disorders) | 0 (0) | 1 (4)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8)
Elevated WBC urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastrointestinal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Headache (General disorders) | 0 (0) | 1 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypercalcemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (6)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (5)
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Hypocalcemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
INR increased (Blood and lymphatic system disorders) | 0 (0) | 1 (9)
Insomnia (General disorders) | 0 (0) | 1 (2)
Lipase increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Musculoskeletal and Connective Tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Nausea (General disorders) | 0 (0) | 1 (3)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Non-cardiac Chest pain (General disorders) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (2)
Platelet Count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Presyncope (General disorders) | 0 (0) | 1 (1)
Sinusitis (General disorders) | 0 (0) | 1 (1)
Skin Biopsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tearing (Ear and labyrinth disorders) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal Spotting (Reproductive system and breast disorders) | 0 (0) | 1 (2)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (7)
Right side chest pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes